CLINICAL TRIAL: NCT00002187
Title: A Randomized Comparison of Two Dosage Schedules of Intravitreal ISIS 2922 for Patients With Advanced Cytomegalovirus Retinitis
Brief Title: A Study of ISIS 2922 in the Treatment of Advanced Cytomegalovirus Retinitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ionis Pharmaceuticals, Inc. (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Model: Parallel | Purpose: Treatment
Other Study IDs: 251D; ISIS 2922-CS9
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1998-12

CONDITIONS: Cytomegalovirus Retinitis; HIV Infections
Keywords: AIDS-Related Opportunistic Infections; Antiviral Agents; Drug Administration Schedule; Cytomegalovirus Retinitis; fomivirsen; Vitreous Body
MeSH Terms: conditions — Cytomegalovirus Retinitis; HIV Infections; AIDS-Related Opportunistic Infections | interventions — fomivirsen

INTERVENTIONS:
Drug: Fomivirsen sodium

SUMMARY:
The purpose of this study is to compare the safety and effectiveness of two dosage schedules for ISIS 2922 in the treatment of advanced cytomegalovirus (CMV) retinitis

DETAILED DESCRIPTION:
This is a multicenter, prospective, randomized, open-label study comparing 2 dosage schedules of ISIS 2922.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Oral ganciclovir.
* Leukocyte growth factors (GM-CSF and G-CSF) for patients with febrile neutropenia.

Patients must have:

* Documented AIDS.
* Clinical diagnosis of advanced CMV retinitis in 1 or both eyes.
* >= 2 previous induction courses with anti-CMV retinitis therapy licensed by a regulatory agency.
* > 25% retinal involvement with CMV retinitis.
* Baseline CMV retinitis lesions which have leading edges > 1000 micrograms from the macula or optic disk.

Prior Medication:

Required:

* >= 2 previous induction courses with anti-CMV retinitis therapy licensed by a regulatory agency.

Allowed:

* All anti-CMV therapies other than ganciclovir must be discontinued no less than 2 days prior to entry.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms and conditions are excluded:

* External ocular infection in the eye to be treated.
* Other herpetic infections of the retina, toxoplasma, retinochoroiditis, or other disease of the fundus that would preclude assessment of CMV retinitis in the eye to be treated.
* Ocular conditions that will obstruct visualization of the posterior ocular structures on the eye to be treated.
* Retinal detachment in the eye to be treated.
* Ganciclovir implant in the eye to be treated.
* Known or suspected allergy to phosphorothioate oligonucleotides or intolerance of ISIS 2922.
* Silicone oil in the eye to be treated.
* Pseudoretinitis pigmentosa.
* Syphilis.

Patients with the following prior conditions are excluded:

* History of surgery to correct retinal detachment in the eye to be treated.
* History of syphilis.

  1. Systemic anti-CMV therapies other than oral ganciclovir.
* Mellaril, Stelazine, chlorpromazine and clofazimine.
* Combination use of ethambutol and fluconazole.
* Investigational medications and/or procedures for the treatment of CMV retinitis in the eye to be treated.
* Ganciclovir implant delivery device in the eye to be treated.
* Ganciclovir other than oral.
* Foscarnet.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (17):
- United States (17):
  - Retina - Vitreous Associates Med Group, Los Angeles, California
  - Community Eye Med Group, Pasadena, California
  - Univ of California San Francisco / SF Gen Hosp, San Francisco, California
  - Dr Jacob Lalezari, San Francisco, California
  - Dr Alan Palestine, Washington D.C., District of Columbia
  - Dr Julio Perez, Fort Lauderdale, Florida
  - Georgia Retina, Atlanta, Georgia
  - Chicago Ctr for Clinical Research, Chicago, Illinois
  - Univ of Illinois, Chicago, Illinois
  - Indiana Univ Med Ctr, Indianapolis, Indiana
  - New York Univ Med Ctr, New York, New York
  - Vitreo - Retinal Consultants, New York, New York
  - Charlotte Eye Ear Nose & Throat Association, Charlotte, North Carolina
  - Duke Univ, Durham, North Carolina
  - Hahnemann Univ Hosp, Philadelphia, Pennsylvania
  - Baylor College of Medicine, Houston, Texas
  - Novum Inc, Seattle, Washington

REFERENCES:
- [Background] New CMV drug won't replace other therapies. AIDS Alert. 1998 Nov;13(11):124-6. PMID 11365968
- [Background] Roehr B. Fomivirsen approved for CMV retinitis. J Int Assoc Physicians AIDS Care. 1998 Oct;4(10):14-6. PMID 11365956